CLINICAL TRIAL: NCT03131778
Title: The Inflammatory Response to Stress and Angiogenesis in Open Versus Laparoscopic Liver Resection for Colorectal Liver Metastases
Brief Title: The Inflammatory Response to Stress and Angiogenesis in Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/048
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Liver Cancer; Colorectal Cancer; Metastatic Cancer; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Liver Resection (Active Comparator): Conventional open liver resection trough subcostal incision
  Interventions: Procedure: Liver resection
- Laparoscopic Liver Resection (Experimental): Pure laparoscopic liver resection without hand assistance
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — liver resections for colorectal liver metastases

SUMMARY:
Patients with resectable liver metastases of colorectal origin will be assigned to laparoscopic liver resection or conventional open liver surgery.

Blood samples will be drawn preoperatively and 24 hours after resection. Determination of Interleukin-6 (IL-6) and IL-8 will be done to assess the stress response between open and laparoscopic liver resection (Elisa test).

The Messenger Ribonucleic Acid (mRNA) of inflammation related factors (cyclooxygenase-2 (COX-2) and Matrix metalloproteinase (MMP-9)), angiogenesis related factor (vascular endothelial growth factor (VEGF) and hypoxia induced factor-1 (HIF-1)) in tumor tissue and normal liver parenchyma will be detected by real-time real time-Polymerase Chain Reaction (RT-PCR).

DETAILED DESCRIPTION:
According to the null hypothesis, no difference in the IL6 postoperative value, between the two groups would be expected. To calculate sample size, a IL6 postoperative value of 100±40 pg/mL in the laparoscopic group and 60±40 mL/m pg/mL in the open group was hypothesized. Considering a two-sided α=0.05 and β=0.1, the minimal sample size required to achieve statistical significance was 17 subjects in both groups in a 1:1 randomization. Laparoscopic group was increased by 20% of patients considering a conversion rate of 20% accordingly. Randomization will be performed using computer-generated random numbers the day before operation and stopped when 20 patients per group will be reached.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Patients with colorectal liver metastases
3. Colorectal liver metastases ≤10 cm in size -

Exclusion Criteria:

1. Patients not fit for laparoscopic surgery due to comorbidities
2. Patients with tumors close or infiltrating the major vessels -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Differences in inflammatory response | Preoperative and postoperative day 1
  Differences in POD 1 levels of IL6 and IL8

SECONDARY OUTCOMES:
Differences in tumor stimulating factors | One week after surgery
  Differences in levels of VEGF, HIF-1α, MMP-9 and COX2 in both humoral and normal liver tissue
Overall Survival | 1-3-5 years
  From surgery to date of death or last follow up. Data will be reported in months
Recurrence free survival | 1-3-5 years
  From surgery to recurrence either in the liver or elsewhere. Data will be reported in months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fretland AA, Sokolov A, Postriganova N, Kazaryan AM, Pischke SE, Nilsson PH, Rognes IN, Bjornbeth BA, Fagerland MW, Mollnes TE, Edwin B. Inflammatory Response After Laparoscopic Versus Open Resection of Colorectal Liver Metastases: Data From the Oslo-CoMet Trial. Medicine (Baltimore). 2015 Oct;94(42):e1786. doi: 10.1097/MD.0000000000001786. PMID 26496309
- [Background] Ueda K, Turner P, Gagner M. Stress response to laparoscopic liver resection. HPB (Oxford). 2004;6(4):247-52. doi: 10.1080/13651820410023987. PMID 18333082
- [Background] Buunen M, Gholghesaei M, Veldkamp R, Meijer DW, Bonjer HJ, Bouvy ND. Stress response to laparoscopic surgery: a review. Surg Endosc. 2004 Jul;18(7):1022-8. doi: 10.1007/s00464-003-9169-7. Epub 2004 May 12. PMID 15136930